CLINICAL TRIAL: NCT05019040
Title: A Phase 1b Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of Multiple Ascending Dose (MAD) of PA1010 Tablets in Chinese Patients With Chronic Hepatitis B Infection
Brief Title: Study of the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of PA1010 in HBV Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Palo Alto Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PA1010-102
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Chronic HBV Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PA1010 5 mg (Experimental): Twelve subjects will be randomly assigned at a 3: 1 ratio to receive either 5 mg of PA1010 tablets or 300 mg of TDF tablets, once daily for 28 days.
  Interventions: Drug: PA1010
- PA1010 10 mg (Experimental): Twelve subjects will be randomly assigned at a 3: 1 ratio to receive either 10 mg of PA1010 tablets or 300 mg of TDF tablets, once daily for 28 days.
  Interventions: Drug: PA1010
- PA1010 20 mg (Experimental): Twelve subjects will be randomly assigned at a 3: 1 ratio to receive either 20 mg of PA1010 tablets or 300 mg of TDF tablets, once daily for 28 days.
  Interventions: Drug: PA1010

INTERVENTIONS:
Drug: PA1010 — TDF as control

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic characteristics of multiple ascending dose (MAD) of PA1010 tablets in Chinese adults with Chronic Hepatitis B.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, controlled, dose-escalation clinical trial, the objective is to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic characteristics of PA1010 tablets in Chinese patients with Chronic Hepatitis B (CHB). There are three dose groups of PA1010 ( 5 mg, 10 mg, and 20 mg) proposed to be tested sequentially in this study. A total of 36 patients with CHB, either hepatitis B e antigen (HBeAg)-positive (+) or HBeAg-negative (-), are planned to be enrolled in this study and will be stratified by HBeAg status by the ratio of 2: 1, that is, 24 of HBeAg + and 12 of HBeAg- patients. Twelve subjects in each dose group were randomly assigned in a 3: 1 ratio to receive either PA1010 tablets or or tenofovir disoproxil fumarate (TDF) tablets. All patients will be dosed for 28 consecutive days, and the dose-related safety, PK, and antiviral efficacy of PA1010 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Sign on the informed consent form to indicate willingness to participate in this study;
2. Male or female CHB patients aged between 18 and 65 (including upper and lower limits), and should meet the following requirements:

   One of the following conditions:
   1. records show that hepatitis B surface antigen (HBsAg) is positive and / or hepatitis B virus deoxyribonucleic acid (HBV DNA) is positive for more than 6 months;
   2. the serum immunoglobulin M (IgM) antibody of HBcAg is negative, and HBsAg is positive;
   3. HBsAg positive and / or HBV DNA positive, and liver biopsy results show chronic hepatitis B (including previous biopsy results);
3. Have not used nucleoside (acid) analogues within 6 months before the first administration, or have received effective, nucleoside(acid) analogues or interferon treatment, but discontinuation of the drug for more than 6 months;
4. For HBeAg positive patients: HBV DNA > 2 × 105 IU/mL； For HBeAg negative patients: HBV DNA > 2 × 104 IU/mL；
5. 1 × Upper limit of normal value (ULN) ≤ alanine aminotransferase (ALT) ≤ 10 × ULN； Serum total bile Hemoglobin ≤ 2 × ULN； Creatinine clearance (clcr) > 70 ml / min (using Cockcroft Gault formula law);
6. Urine protein is negative or 1+ (it is necessary to add 24 hours of urine protein quantification when 1+. If within the normal range, selected);
7. No major disease history, and the physical examination, vital signs, 12 lead electrocardiogram (ECG) and laboratory examination results are normal during the screening period , although they exceed the normal reference value range, they are judged by the investigator to be of no clinical significance;
8. Subjects are forbidden to donate blood or use drugs within 30 days after the last dose;
9. During the study period (from signing the informed consent to the last follow-up) and within 6 months after the last dose, sperm donation and egg donation are prohibited, and there is no possibility of pregnancy (or sexual partner pregnancy), childbirth and lactation, at least one of the following conditions is met:

   1. Menopausal women who have menopause for more than 12 months or undergo sterilization (such as hysterectomy, ligation of both fallopian tubes or bilateral ovariectomy);
   2. For premenopausal women, pregnancy tests in the screening period and baseline period are negative, and they are willing to take more than one effective contraceptive method from the screening period to 6 months after the last dose, including intrauterine device, tubal ligation, double barrier method (condom / vaginal diaphragm + spermicide) and male partner vas deferens ligation, but excluding oral contraceptives;
   3. Men are willing to take more than one effective contraceptive method within 6 months after the last dose, including vasectomy, double barrier method, female partner's use of contraceptives, intrauterine device or tubal ligation, etc;
   4. Avoid sexual life within 6 months after the last dose;
10. Be able to communicate with clinical staff and comply with the requirements of this study.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from the study:

1. There are any medical conditions that the investigator believes may increase the risk of subjects participating in the study (especially the history of esophageal or gastrointestinal ulcer), may interfere with the absorption, distribution, metabolism or excretion of drugs, or may weaken the compliance with the study protocol;
2. Patients with liver diseases other than hepatitis B, including but not limited to patients with chronic alcoholic hepatitis, drug-induced liver injury, autoimmune liver disease, known Gilbert syndrome and other hereditary liver diseases;
3. Any history or current signs of liver decompensation (ascites, hepatic encephalopathy or esophageal and gastric varices bleeding) at any time before or at the time of screening, child Pugh grade B or C;
4. Those who have received solid organ or bone marrow transplantation;
5. History of severe kidney disease (judged by the researcher) or current signs;
6. Serious bone diseases (such as osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, chondrosis) or multiple bone diseases fold;
7. Liver malignant tumor or other untreated malignant tumor was diagnosed before the first administration ;
8. Have received any other study drug within 90 days before the first dose;
9. Those who have used other nucleosides (acids) or interferons within 6 months before the first administration;
10. Before the first administration, stop the prescription drug or over-the-counter drug that other researchers believe will affect the evaluation results of this study less than 14 days or 5 half lives of the drug (whichever is longer);
11. Blood donation or massive blood loss (>400 ml) within 3 months before the first administration of the study drug;
12. Major surgery or trauma within 6 months before the first administration;
13. Take drinks or food containing grapefruit, pomegranate, papaya, grape and carambola within 14 days before the first administration, or disagree to avoid taking any drinks or food containing grapefruit, pomegranate, papaya, grape and carambola every day during the test;
14. Have taken any food or drink rich in caffeine and xanthine (coffee, tea, coke, chocolate, seafood, animal liver, etc.) within 48 hours before the first administration, or do not agree to avoid taking any food or drink rich in caffeine and xanthine (coffee, tea, coke, chocolate, seafood, animal liver, etc.) every day during the test;
15. Abnormal ECG in screening or baseline period, which is judged to be clinically significant by the investigator; Or QTCF > 450 ms in screening or baseline period;
16. Have a history of heart disease, including a family history of sudden death caused by cardiac causes or QT interval prolongation syndrome;
17. Difficulty in venous blood collection, or known to have a history of needle fainting and blood fainting for many times;
18. Clinical or laboratory evidence shows that: hepatitis C virus (HCV), hepatitis D disease (HDV) persons carrying / infected with Treponema pallidum (TP) or human immunodeficiency virus (HIV);
19. Known to have a history of allergy to the study drug and its excipients;
20. Any history of drug abuse or urine drug test (+) during screening period;
21. Have a regular drinking history within 6 months before screening. Women have more than 7 cups / week, men have more than 14 cups / week (1 cup =5 ounces of wine or 12 ounces of beer or 1.5 ounces of spirits) or the alcohol test exceeds the standard during the screening period;
22. Smokers (smoking 10 or more cigarettes a day).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Evaluation the change from baseline in Serum HBV DNA in patients | 28 days
  The primary efficacy endpoint is the change from baseline in Serum HBV DNA in patients on day 28 in all patients. The safety and tolerance are also observed in all treatment groups.
Evaluation the rate of change from Baseline in Serum HBV DNA | 28 days
  Rate of change from Baseline in Serum HBV DNA
Evaluation the change from Baseline in Serum HBsAg | 28 days
  Change from Baseline in Serum HBsAg
Evaluation the change from Baseline in Serum ALT | 28 days
  Change from Baseline in Serum ALT
Number of subjects experiencing adverse events (AEs) | 28 days
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical study subject administered a medicinal product which does not necessarily have a causal relationship with this treatment.
Pharmacokinetics of single dose of PA1010-Cmax | 28 days
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Maximum Observed Plasma Concentration (Cmax)
Pharmacokinetics of single dose of PA1010-Tmax | 28 days
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Time to Reach Maximum Observed Plasma Concentration (Tmax)
Pharmacokinetics of single dose of PA1010-AUC | 28 days
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Area Under the Plasma Concentration-Time Curve (AUC)
ECG parameter-QTc interval、PR interval、QRS duration | 28 days
  A 12 lead electrocardiogram (ECG) will be recorded using an ECG machine that automatically measures QTc interval、PR interval、QRS duration
Number of new abnormal signs with clinical significance | 28 days
  Physical examination records include: skin, lymph nodes, head and neck (including thyroid), nervous system examination (including but not limited to speech, cranial nerves, motor ability, tendon reflex, sensation, ataxia), chest (heart, lung), abdomen (liver, gallbladder, spleen, kidney), etc.
Body temperature, blood pressure, pulse, respiratory rate | 28 days
  Vital signs body temperature, blood pressure, pulse, respiratory rate

SECONDARY OUTCOMES:
Pharmacokinetics of single dose of PA1010-T1/2 | 28 days
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Elimination Half-Life Period (T1/2）
Pharmacokinetics of single dose of PA1010-Vz/F | 28 days
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Apparent Volume of Distribution(Vz/F)
Pharmacokinetics of single dose of PA1010-CL/F | 28 days
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Apparent Clearance(CL/F)
Pharmacokinetics of single dose of PA1010-λz | 28 days
  Blood samples will be collected serially, and the concentrations of PA1010 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Elimination Rate Constant(λz)

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, MD, Principal Investigator — Beijing Tsinghua Changgung Hospital affiliated to Tsinghua University
Locations (4):
- China (4):
  - Beijing Tsinghua Changgung Hospital affiliated to Tsinghua, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Southern Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No